CLINICAL TRIAL: NCT01168622
Title: Impact of Race/Ethnicity on Platelet Function
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0144-10-EP
Record Dates: First submitted 2010-06-25; First posted 2010-07-23 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood or saliva samples will be collected for DNA extraction and genotyping of CYP2C19 and other relevant genes.
Oversight: Data Monitoring Committee: No

SUMMARY:
The effects of race/ethnicity on platelet function and response to antiplatelet agents will be assessed using healthy participants and coronary heart disease patients from at least 5 racial/ethnic groups.

DETAILED DESCRIPTION:
The effects of race/ethnicity on platelet function and response to antiplatelet agents will be assessed using 125 healthy subjects, 250 coronary heart disease patients treated with aspirin, and 250 coronary heart disease patients treated with aspirin and a P2Y12 receptor antagonist, clopidogrel or prasugrel. A minimum of 25 healthy people, 50 people taking only aspirin, and 50 people taking aspirin and clopidogrel/prasugrel will be recruited for at least 5 racial/ethnic groups.

ELIGIBILITY:
Inclusion Criteria: Each subject must fulfill the following criteria in order to be included in the study.

* The subject must be capable of understanding the nature of the study and executing an informed consent document.
* The subject must be aged 19 years or older.
* For healthy subjects, the subject must deny taking any medications that affect platelet function for at least 7 days before blood collection.
* For diseased patients, subjects with documented CAD are eligible to participate if they have been treated with antiplatelet therapy of aspirin (81 to 325 mg/day) with and without clopidogrel (75 mg/day) or another P2Y12 antagonist for at least one month.

Exclusion Criteria: For healthy volunteers, subjects who fulfill one or more of the following criteria will be excluded from the study.

* taking medications for chronic cardiovascular diseases.
* illnesses requiring hospitalization or surgery within the last three months.
* history of drug or alcohol abuse.
* history of recent anemia or thrombocytopenia.
* history of excessive bleeding or thrombosis.
* pregnancy.

For coronary heart disease subjects, subjects who fulfill one or more of the following criteria will be excluded from the study.

* illnesses requiring hospitalization or surgery within the last one month.
* history of drug or alcohol abuse.
* history of recent anemia or thrombocytopenia.
* pregnancy.
* recent bleeding diathesis
* malignancy
* renal insufficiency
* liver dysfunction
* treatment with warfarin or glycoprotein (GP) IIb/IIIa antagonists during the preceding 14 days

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy people and coronary heart disease patients taking aspirin or aspirin and clopidogrel or prasugrel
Sampling Method: Non-Probability Sample
Enrollment: 625 (Estimated)
Dates: Start 2010-06-01 (Actual); Primary Completion 2013-03-30 (Actual); Study Completion 2013-03-30 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity | baseline only
  Platelet reactivity as measured by platelet function tests

CONTACTS AND LOCATIONS:
Overall Officials: Julie H Oestreich, PharmD, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States